CLINICAL TRIAL: NCT05805280
Title: IntravasCular Imaging-Guided Versus AngiogRaphy-GUided Drug-Eluting Stent Implantation for Fermoropopliteal Artery Disease (ICARUS Trial); A Feasibility Study
Brief Title: IntravasCular Imaging-Guided Versus AngiogRaphy-GUided Drug-Eluting Stent Implantation for Fermoropopliteal Artery Disease
Acronym: ICARUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Seung-Whan Lee, M.D., Ph.D., Part of cardiology, Principal Investigator, associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1514
Record Dates: First submitted 2023-03-22; First posted 2023-04-07 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Femoropopliteal Disease

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomized at a ratio 1:1 to two treatment arms by a computer-generated randomization sequence with a permutated block size 4.
  a) intravascular ultrasound-guided group or b) Angiography-guided group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravascular ultrasound-guided group (Experimental): In the intravascular ultrasound-guided group, intravascular ultrasound will be either automatically (1 mm/sec) or manually (5-10 mm/sec) pulled back at a constant speed according to the lesion length. Stent size and length are selected by information acquired from on-line intravascular ultrasound examination, and adjunct high-pressure dilation is performed to achieve stent optimization based on the intravascular ultrasound finding
  Interventions: Device: intravascular ultrasound-guided group
- angiography-guided group (Active Comparator): In the angiography-guided group, stent size and length are chosen by visual estimation, and adjunctive high-pressure dilation is performed if an optimal result, defined as angiographic residual diameter stenosis of less than 30% by visual estimation and the absence of angiographically detected dissection, , was not achieved
  Interventions: Device: angiography-guided group

INTERVENTIONS:
Device: intravascular ultrasound-guided group — intravascular ultrasound use
  Arms: intravascular ultrasound-guided group
Device: angiography-guided group — angiography-guided use
  Arms: angiography-guided group

SUMMARY:
Objectives: 1) To evaluate the feasibility of using intravascular ultrasound to assess lesion morphology, select an appropriate stent size and landing zone 2) To compare the primary patency rates after intra vascular imaging-guided versus angiography-guided stent implantation for the treatment of fermoropopliteal artery segment lesions.

Hypothesis: One of the key determinants of the device failure is inappropriate landing zone, selection of smaller stent relative to the reference vessel diameter, and lack of high-pressure post-dilatation in a necessary post-stent segment. Therefore, intravascular ultrasound-guided selection of appropriate landing zone, stent size and balloon size for high pressure post-dilation may maximize the benefits of stent use and improve patency duration. the investigators hypothesize that intravascular ultrasound-guided stent implantation is superior to angiography-guided stent implantation with respect to 12 months primary patency in patients with significant femoropopliteal disease

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized comparison feasibility trial involving patients with significant femoropopliteal disease who are undergoing drug-eluting stent (paclitaxel-eluting, durable-polymer-coated Eluvia stent) implantation. Patients with symptoms attributable to limb ischemia are eligible for enrollment if the culprit lesions are suitable for stent implantation based on angiographic findings. The detailed information for inclusion and exclusion criteria is described below in session 7. Patients meeting inclusion criteria without any exclusion criteria will be randomized to either intravascular ultrasound-guided or angiography-guided group immediately before the endovascular intervention. In the intravascular ultrasound-guided group, intravascular ultrasound will be either automatically (1 mm/sec) or manually (5-10 mm/sec) pulled back at a constant speed according to the lesion length. Stent size and length are selected by information acquired from on-line intravascular ultrasound examination, and adjunct high-pressure dilation is performed to achieve stent optimization based on the intravascular ultrasound finding. For the selection of the landing zone and stent length, intravascular ultrasound and fluoroscopy images should be recorded simultaneously to link intravascular ultrasound images with location preferably using a ruler. For the selection of stent size and assessment of stent optimization, external elastic membrane area (EEM) before ballooning and minimal stent area (MSA) (i.e, the smallest cross-sectional area within the stent) after post-dilation are assessed. intravascular ultrasound is used at any step of the procedure before, during, or after stenting. However, image examination is mandatory before and after stenting. In the angiography-guided group, stent size and length are chosen by visual estimation, and adjunctive high-pressure dilation is performed if an optimal result, defined as angiographic residual diameter stenosis of less than 30% by visual estimation and the absence of angiographically detected dissection, was not achieved. Stent size is chosen at the operator's discretion in both groups, with diameters 1 or 2 mm larger than the reference diameter assessed either by intravascular ultrasound or visual estimation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 20 years up to 85 years of age
* Intermittent claudication or tissue loss suitable for elective endovascular intervention (Rutherford category 2,3,4, or 5)
* Significant native superficial femoral or proximal popliteal artery lesions suitable for stent implantation. Restenotic lesions can be enrolled at least 12-month after the index procedure uding plain balloon or drug-coated balloon.
* Total lesion length of 30 to 220 mm
* Reference vessel diameter of 4 - 6 mm
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Existence of a stent in the target vessel
* Previous use of atherectomy device in the target vessel
* Use of drug-coated balloon in the target vessel within 12-month
* Untreatable significant stenosis or occlusion (diameter stenosis ≥70%) in all 3 infrapopliteal arteries (patient can be enrolled if at least 1 patent outflow artery to the ankle (diameter stenosis <50%) can be achieved by treatment during the index procedure)
* A known intolerance or contraindication to antiplatelet drugs (aspirin or clopidogrel)
* Unwillingness or inability to comply with the procedures described in this protocol.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
patency at 12 months after treatment | 12 month after randomization
  peak systolic velocity ratio 2.4 or lower as assessed by the duplex ultrasound, in the absence of clinically driven target lesion revascularization or bypass of the target lesion.
Number of procedure related death | 30 Days post procedure
  procedure related death through 30 days post-procedure
Number of major amputation of the target limb or target-lesion revascularization | 12 month after randomization
  major amputation of the target limb through 12 months, or target-lesion revascularization through 12 months

SECONDARY OUTCOMES:
technical success | within 24 hours
  deployment of the stent to the target lesion to achieve residual angiographic stenosis ≤30%
procedural success | within 24 hours
  technical success without major adverse events
Rutherford category score | 12 month after randomization
  1. Stage 0 - Asymptomatic
  2. Stage 1 - Mild claudication
  3. Stage 2 - Moderate claudication
  4. Stage 3 - Severe claudication
  5. Stage 4 - Rest pain
  6. Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot
  7. Stage 6 - Severe ischemic ulcers or frank gangrene

CONTACTS AND LOCATIONS:
Overall Officials: Pil Hyung Lee, MD, Principal Investigator — Asan Medical Center
Locations (8):
- South Korea (8):
  - Inje University Busan Paik Hospital, Busan
  - Veterans Hospital, Daegu
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Severance Cardiovascular Hospital, Seoul
  - Veterans Health Service Medical Center, Seoul
  - Ajou University Medical Center, Suwon

IPD SHARING:
Plan to Share IPD: No